CLINICAL TRIAL: NCT00181727
Title: Open-Label Study of Divalproex Sodium Extended Release for the Treatment of Mania in Children Ages 6-12 With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Study of Depakote ER for the Treatment of Mania in Children Ages 6-12 With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD; Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-001557
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar Disorder; Mania
Keywords: bipolar disorder; mania; depakote ER; children
MeSH Terms: conditions — Bipolar Disorder; Mania

INTERVENTIONS:
Drug: divalproex sodium extended release

SUMMARY:
This is an open-labeled study of Divalproex Sodium Extended Release (Depakote ER), testing its efficacy for the treatment of mania in children between the ages of 6-12 who have been diagnosed with Bipolar I, Bipolar II, and Bipolar Spectrum Disorders. This is an exploratory, pilot study, seeking to determine whether Divalproex Sodium Extended Release is efficacious and well tolerated in the treatment of youth with pediatric bipolar and bipolar spectrum disorder, and the study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

DETAILED DESCRIPTION:
Initial clinical evidence suggests that Divalproex Sodium may play a therapeutic role in the management of pediatric bipolar disorder. Its new Extended Release formulation offers the advantage of once a day dosing. Although the precise mechanisms by which Divalproex Sodium exerts its therapeutic effects remains unknown, it has been suggested that its activity may be related to increased brain concentrations of gamma-aminobutyric acid (GABA). Although the shorter acting formulation Divalproex Sodium is FDA approved for the treatment of adult bipolar disorder, its Extended Release formulation is currently only FDA approved for adults for the prophylactic treatment of migraine headaches and has not yet been studied in patients with mania. Three studies of Divalproex Sodium have documented safety and efficacy of this compound, as well as superiority over placebo, in the treatment of adults with bipolar disorder.

This medication has not, however, been adequately investigated in children. The proposed study includes 1) an 8-week acute period, during which participants are observed during weekly visits, and up to an 8-month extension period, during which participants see a study clinician on a monthly basis, to document the response rate 2) assessment of the impact of Divalproex Sodium Extended Release on functional capacities (quality of life, psychosocial function) and cognition, 3) careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 6-12 years of age.
2. Subjects must have a DSM-IV diagnosis of bipolar I, bipolar II disorder or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders and Schizophrenia Epidemiological Version)(Kaufman, Birmaher et al. 1997). Bipolar spectrum disorder (or sub-threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but meet fewer elements in criteria B (only require 2 items for elation category and 3 for irritability).
3. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
4. Subjects and their legal representative must be considered reliable.
5. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
6. Subjects must have an initial score on the Y-MRS total score of at least 20.
7. Subject must be able to participate in mandatory blood draws.
8. Subject must be able to swallow pills.
9. Subjects with comorbid ADHD, ODD, CD, anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of the exclusionary criteria.
10. For concomitant stimulant therapy used to treat ADHD, subjects must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the stimulant therapy will not change throughout the duration of the initial phase of the study.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Uncorrected hypothyroidism or hyperthyroidism.
4. History of severe allergies or multiple adverse drug reactions.
5. Non-febrile seizures without a clear and resolved etiology.
6. Leukopenia or history of leukopenia without a clear and resolved etiology.
7. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months.
8. Judged clinically to be at serious suicidal risk.
9. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
10. A non-responder or a history of intolerance to Divalproex Sodium Extended Release to an adequate trial (2 months or more at an adequate dose) as determined by the clinician.
11. Receiving treatment with Strattera.
12. Current diagnosis of schizophrenia.
13. Pregnant or nursing females.
14. Non English speaking subjects will not be allowed into the study for the following reasons: a) the assessment instruments are not available and have not been adequately standardized in other languages; b) our clinical trials facility is located in Cambridge and not in the MGH main campus without the availability of translators; c) psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes:
Scores on the Young Mania Rating Scales, two subscales of the MRS:
1) the Manic Syndrome Scale (MSS)
2) the Behavior and Ideation Scale (BIS)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States